CLINICAL TRIAL: NCT00477607
Title: Prevention of Cisplatin Ototoxicity With the Antioxidant Alpha-Lipoic Acid
Brief Title: Alpha-Lipoic Acid in Preventing Hearing Loss in Cancer Patients Undergoing Treatment With Cisplatin
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Collaborators: Oregon Health and Science University (Other)
Responsible Party: Sponsor
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: C4697-R; CDR0000546570 (Other Grant/Funding Number: VA RR&D); NCRAR-VA-1810 (Other Grant/Funding Number: VA RR&D); OHSU-3288 (Other Grant/Funding Number: VA RR&D); NCT00570596 (obsolete NCT alias)
Record Dates: First submitted 2007-05-23; First posted 2007-05-24 (Estimated); Results first posted 2014-01-29 (Estimated); Last update posted 2014-03-07 (Estimated); Status verified 2014-02

CONDITIONS: Ototoxicity; Unspecified Adult Solid Tumor
MeSH Terms: conditions — Ototoxicity | interventions — Thioctic Acid

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm 1 (Experimental): Receiving alpha-lipoic acid during cisplatin treatment.
  Interventions: Drug: alpha-lipoic acid; Behavioral: Audiology; Biological: laboratory biomarker analysis
- Arm 2 (Placebo Comparator): Receiving placebo during cisplatin treatment
  Interventions: Behavioral: Audiology; Biological: laboratory biomarker analysis; Drug: Placebo

INTERVENTIONS:
Drug: alpha-lipoic acid — Supplements (1200mg once a day) or placebo will be administered to each patient prior to first cisplatin treatment and continue until 3 months after last treatment.
  Other Names: lipoic acid
  Arms: Arm 1
Behavioral: Audiology — otoscopy, immittance screening, noise exposure questionnaire and individualized behavioral pure-tone in the convention and high-frequency ranges.
  Other Names: ototoxicity monitoring
Biological: laboratory biomarker analysis — Plasma concentrations of Malondialdehyde (MDA) will be measures as an indicator of oxidative stress.
  Other Names: MDA
Drug: Placebo — Placebo will be administered to each patient prior to first cisplatin treatment and continue until 3 months after last treatment.
  Arms: Arm 2

SUMMARY:
RATIONALE: Alpha-lipoic acid may prevent or lessen hearing loss caused by cisplatin.

PURPOSE: This randomized clinical trial is studying the effectiveness of alpha-lipoic acid in preventing hearing loss in cancer patients undergoing treatment with cisplatin.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

Determine the ability of alpha-lipoic acid supplementation to prevent or reduce the incidence and severity of hearing loss in cancer patients undergoing treatment with cisplatin.

Secondary

Determine if this drug improves the oxidative state, as measured by a malondialdehyde measurement of oxidative stress, thereby protecting the patient against ototoxic-induced hearing loss.

OUTLINE: This is a placebo-controlled, double-blind, randomized, multicenter study. Patients are stratified by cancer stage and institution. Patients are randomized to 1 of 2 treatment arms.

Arm I: Patients receive oral alpha-lipoic acid supplement once a day beginning 1 week before the start of cisplatin treatment and continuing for up to 1 month after the completion of cisplatin. During cisplatin treatment, patients discontinue supplement 1 day prior to the cisplatin treatment and resume daily supplements 2 days post treatment.

Arm II: Patients receive oral placebo supplement once a day beginning 1 week before the start of cisplatin and continuing for up to 1 month after the completion of cisplatin. During cisplatin treatment, patients discontinue supplement 1 day prior to the cisplatin treatment and resume daily supplements 2 days post treatment.

Hearing and ototoxicity are assessed at baseline, on each day of chemotherapy, and at 1 and 3 months post chemotherapy.

Blood samples are collected periodically to measure malondialdehyde and alpha-lipoic acid levels.

After completion of treatment with cisplatin, patients are followed for 3 months.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of cancer
* Receiving therapeutic treatment with cisplatin
* Fertile patients must use effective contraception during and for 3 months after completion of study treatment
* Cognitively and physically able to participate in the study
* Must be able to provide reliable behavioral threshold responses (patient must meet intra-session reliability criterion of +/- 5 dB)
* At least 6 months since prior treatment with cisplatin or other ototoxic medications (e.g., aminoglycoside antibiotics)
* At least 6 months since prior and no concurrent radiotherapy for head and neck tumors
* Concurrent radiotherapy targeted below the neck allowed
* More than 1 month since prior alpha-lipoic acid supplements

Exclusion Criteria:

* No aggressive behavior as indicated in electronic chart notes
* No documented dementia
* No Alzheimer's disease
* No severe psychosocial disorder
* No active or recent history of middle ear disorder based on otoscopy, tympanometry, immittance, or notes in patient chart
* No renal disease
* No Meniere's disease or retrocochlear disorder based on patient report or notes in patient's chart
* Not receiving treatment for diabetes mellitus
* No concurrent vincristine or vinblastine
* No other concurrent investigational therapy
* No other concurrent antioxidants or vitamin E > 100 IU per day

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2007-10; Primary Completion 2011-03 (Actual); Study Completion 2011-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dawn L Martin, Principal Investigator — Portland VA Medical Center, Portland, OR
Locations (2):
- United States (2):
  - VA Medical Center, Portland, Portland, Oregon
  - Oregon Health & Science University, Portland, Oregon

RESULTS

PARTICIPANT FLOW:
Groups:
- Alpha-lipoic Acid: Receiving alpha-lipoic acid during cisplatin treatment.
  alpha-lipoic acid : Supplements (1200mg once a day) was administered to each patient prior to first cisplatin treatment and continued until 3 months after last treatment.
- Placebo: Receiving placebo during cisplatin treatment
  Placebo supplements (1200mg once a day) were administered to each patient prior to first cisplatin treatment and continued until 3 months after last treatment.
Period: Overall Study
Arm/Group | Alpha-lipoic Acid | Placebo
Started | 19 | 20
Completed | 12 | 13
Not Completed | 7 | 7
Not completed — Lost to Follow-up | 7 | 7

BASELINE CHARACTERISTICS:
Groups:
- Arm 1: Receiving alpha-lipoic acid during cisplatin treatment.
  laboratory biomarker analysis : Plasma concentrations of Malondialdehyde (MDA) will be measures as an indicator of oxidative stress.
  alpha-lipoic acid : Supplements (1200mg once a day) or placebo will be administered to each patient prior to first cisplatin treatment and continue until 3 months after last treatment.
  Audiology : otoscopy, immittance screening, noise exposure questionnaire and individualized behavioral pure-tone in the convention and high-frequency ranges.
- Arm 2: Receiving placebo during cisplatin treatment
  Audiology : otoscopy, immittance screening, noise exposure questionnaire and individualized behavioral pure-tone in the convention and high-frequency ranges.
  alpha-lipoic acid : Supplements (1200mg once a day) or placebo will be administered to each patient prior to first cisplatin treatment and continue until 3 months after last treatment.
  laboratory biomarker analysis : Plasma concentrations of Malondialdehyde (MDA) will be measures as an indicator of oxidative stress.
- Total: Total of all reporting groups
Arm/Group | Arm 1 | Arm 2 | Total
Number analyzed (Participants) | 19 | 20 | 39
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 12 | 15 | 27
  >=65 years | 7 | 5 | 12
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.0 (10.2) | 60.6 (12.3) | 61.2 (11.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 1 | 1
  Male | 19 | 19 | 38
Region of Enrollment [Number; unit: participants]
  United States | 19 | 20 | 39

OUTCOME MEASURES:

1. Primary Outcome: Ototoxicity Measurement
Description: Any American Speech and Hearing Association (ASHA)-significant hearing loss in the Sensitive Region for Ototoxicity frequencies between baseline measurement and any follow-up measurement.
  ASHA criteria are defined as
  * 20 decibel (dB) increase at any test frequency,
  * 10 dB increase at any two consecutive test frequencies, or loss of response where there was previously a response at any three test frequencies.
Time Frame: Baseline measurement occurred prior to first cisplatin treatment session. Follow-up measurements occurred up to 3 months after last cisplatin treatment.
Population: Intent-to-treat (ITT)
Measure: Number; unit: participants
Arm/Group | Arm 1 | Arm 2
Number analyzed (Participants) | 10 | 13
participants | 7 | 7
Statistical Analysis 1: Comparison: Arm 1 vs Arm 2; H0: pr(Hearing loss arm 1) = pr(Hearing loss arm 2); Test type: Superiority or Other; p = 0.89, Fisher Exact; No adjustments. Right one-sided p-value; Odds Ratio (OR) = 2, 95% CI 2-sided [0.4 to 11.4]

2. Secondary Outcome: Malondialdehyde (MDA) Levels
Description: Computed maximum increase relative to baseline for each subject = (max MDA during treatment) - baseline MDA level.
Time Frame: as for outcome 1
Population: Non-missing MDA measurements from 23 subjects in primary outcome analysis
Measure: Mean (Standard Deviation); unit: uM=micro-moles/liter
Arm/Group | Arm 1 | Arm 2
Number analyzed (Participants) | 10 | 11
uM=micro-moles/liter | 0.27 (1.00) | 0.47 (0.83)
Statistical Analysis 1: Comparison: Arm 1 vs Arm 2; H0: mean (MDA arm 1) = mean (MDA Arm 2); Test type: Superiority or Other; p = 0.63, t-test, 2 sided; Mean Difference (Final Values) = -0.195, 95% CI 2-sided [-1.03 to 0.64], Standard Error of Mean 0.3999

3. Secondary Outcome: Total Amount of Prescribed Cisplatin Dose Administered
Description: Maximum cumulative dose of cisplatin (mg/m^2) administered during the course of chemotherapy.
Time Frame: cisplatin treatment period between 10 weeks and up to 16 weeks.
Population: Subjects from the original 39 recruited who had sufficient chemotherapy data recorded to measure cumulative dose.
Measure: Mean (Standard Deviation); unit: mg/m^2
Arm/Group | Arm 1 | Arm 2
Number analyzed (Participants) | 19 | 20
mg/m^2 | 239.7 (92.6) | 191.5 (110.5)
Statistical Analysis 1: Comparison: Arm 1 vs Arm 2; H0: mean(max dose arm 1) = mean(max dose arm 2); Test type: Superiority or Other; p = 0.15, t-test, 2 sided; Mean Difference (Final Values) = 48.2, 95% CI 2-sided [-18.1 to 114.6], Standard Error of Mean 32.7

ADVERSE EVENTS:
Arm/Group | Arm 1 | Arm 2
Serious Adverse Events (participants affected / at risk) | 5/19 | 6/20
Other Adverse Events (participants affected / at risk) | 3/19 | 2/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm 1 (N=19) | Arm 2 (N=20)
Neutropenia (Blood and lymphatic system disorders) | 1 (1) | 2 (2)
Nausea/vomitting (Gastrointestinal disorders) | 1 (1) | 0 (0)
Blood transfusion (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Acute Renal Failure (Renal and urinary disorders) | 0 (0) | 3 (3)
Pancreatitis (Endocrine disorders) | 0 (0) | 1 (1)
Esophagitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
sceptic shock (Infections and infestations) | 1 (1) | 0 (0)
hypoxic respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm 1 (N=19) | Arm 2 (N=20)
Small bowel obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1)
Spine pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Distended abdomen (Gastrointestinal disorders) | 1 (1) | 0 (0)
Atrial Fibrillation (Cardiac disorders) | 1 (1) | 0 (0)
Muscle Weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
Missing data constraints have the number of subjects in the study being different for different outcomes.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No